CLINICAL TRIAL: NCT02821000
Title: A Phase Ib Study of Pembrolizumab (MK-3475) in Chinese Subjects With Locally Advanced or Metastatic Melanoma (Keynote-151)
Brief Title: Safety and Efficacy Study of Pembrolizumab (MK-3475) in Chinese Participants With Locally Advanced or Metastatic Melanoma (MK-3475-151/KEYNOTE-151)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3475-151; MK-3475-151 (Other: Merck Protocol Number); KEYNOTE-151 (Other: Merck)
Record Dates: First submitted 2016-06-29; First posted 2016-07-01 (Estimated); Results first posted 2019-03-21 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2023-12

CONDITIONS: Melanoma
Keywords: PD1; PD-1; PDL1; PD-L1
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pembrolizumab (Experimental): Participants receive pembrolizumab 2 mg/kg intravenously on Day 1 of each 3-week cycle for up to 35 administrations (up to approximately 2 years).
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — Intravenous infusion
  Other Names: MK-3475

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and objective response rate (ORR) of pembrolizumab (MK-3475) in Chinese participants with locally advanced or metastatic melanoma, with disease progression following first line chemotherapy or targeted therapy. ORR will be based on Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1).

With Amendment 6 (effective date 18-Mar-2022), once the study objectives have been met or the study has ended, participants will be discontinued from this study and may be enrolled in an extension study to continue protocol-defined assessments and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Is of the Chinese descent, was born in China, and has a Chinese home address.
* Has histologically confirmed diagnosis of locally advanced (unresectable Stage III) or metastatic (Stage IV) melanoma not amenable to local therapy.
* Participant may not have a diagnosis of uveal or ocular melanoma.
* Overall proportion of participants with mucosa melanoma will be no more than 22%.
* Has failed the first line chemotherapy (excluding adjuvant or neoadjuvant therapy) or targeted therapy for melanoma.
* Has at least one measurable lesion as defined by RECIST 1.1 on imaging studies (computed tomography [CT] or magnetic resonance imaging [MRI]).
* Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Has an anticipated life expectancy of at least 3 months.
* Demonstrates adequate organ function.
* Has provided tissue for anti-programmed cell death ligand-1 (PD-L1) expression evaluation from an archival tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated.
* Has documented BRAF mutation status or is willing to provide a tumor tissue for BRAF genotyping.
* Females may be enrolled in the study if they are:
* Of non-childbearing potential which is defined as:

  * Is ≥45 years of age and has not had menses for greater than 2 years.
  * Is amenorrheic for <2 years without a hysterectomy and oophorectomy and has a follicle stimulating hormone (FSH) value in the postmenopausal range upon screening evaluation, and/or,
  * Is status post hysterectomy, oophorectomy or tubal ligation.
* Female and male participants of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study treatment. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the participant.

Exclusion Criteria:

* Has received prior therapy with an anti-programmed cell death 1 (anti-PD-1), anti-PD-L1, anti-PD-L2 agents.
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigation device within 4 weeks of the first dose of study drug.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to the first dose of study drug or who has not recovered (i.e., ≤ Grade 1 or baseline) from AEs due to agents administered more than 4 weeks earlier.
* Has had chemotherapy, targeted small molecule therapy, radiotherapy within 2 weeks prior to the first dose of study drug, or who has not recovered (i.e., ≤ Grade 1 or baseline) from AEs due to a previously administered agent.
* Has a known history of another (including unknown primary) malignancy within 5 years prior to first dose of study drug. (Exceptions include adequately treated Stage 1 or Stage 2 basal/squamous cell carcinoma of the skin, superficial bladder cancer, or cancer in situ which has undergone potentially curative therapy.)
* Is expected to require any other form of systemic or localized antineoplastic therapy while in study.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs).
* Is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 1 week prior to the first dose of study drug.
* Has an active infection requiring intravenous systemic therapy.
* Has received a live vaccine within 4 weeks prior to the first dose of study drug.
* Has a known hypersensitivity to the components of the study drug or another mAb.
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Is known to be Human Immunodeficiency Virus (HIV) positive.
* Has known active Hepatitis B or C.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit (Visit 1) through 120 days after the last dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2016-07-08 (Actual); Primary Completion 2017-12-27 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Si L, Zhang X, Shu Y, Pan H, Wu D, Liu J, Lou F, Mao L, Wang X, Wen X, Gu Y, Zhu L, Lan S, Cai X, Diede SJ, Zhou Y, Ge J, Li J, Wu H, Guo J. A Phase Ib Study of Pembrolizumab as Second-Line Therapy for Chinese Patients With Advanced or Metastatic Melanoma (KEYNOTE-151). Transl Oncol. 2019 Jun;12(6):828-835. doi: 10.1016/j.tranon.2019.02.007. Epub 2019 Apr 10. PMID 30981094
- [Derived] Si L, Zhang X, Shu Y, Pan H, Wu D, Liu J, Mao L, Wang X, Wen X, Gu Y, Zhu L, Lan S, Cai X, Diede SJ, Dai H, Niu C, Li J, Guo J. Pembrolizumab in Chinese patients with advanced melanoma: 3-year follow-up of the KEYNOTE-151 study. Front Immunol. 2022 Oct 11;13:882471. doi: 10.3389/fimmu.2022.882471. eCollection 2022. PMID 36304457
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab: Participants received pembrolizumab 2 mg/kg intravenous (IV) on Day 1 of each 21-day cycle. Eligible participants received up to 17 additional administrations (up to approximately 1 year) of pembrolizumab 2 mg/kg on day 1 of each 21-day cycle.
Period: Overall Study
Arm/Group | Pembrolizumab
Started | 103
Treated | 103
Completed | 0
Not Completed | 103
Not completed — Death | 89
Not completed — Sponsor Decision | 12
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 103
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: All enrolled participants
  Years | 50.5 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All enrolled participants
  Participants
    Female | 59
    Male | 44
Race (NIH/OMB) [Count of Participants; unit: Participants] — The race of participants is presented. Population: All enrolled participants
  Participants
    American Indian or Alaska Native | 0
    Asian | 103
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 0
    More than one race | 0
    Unknown or Not Reported | 0
Programmed Cell Death-Ligand 1 (PD-L1) Expression Status [Count of Participants; unit: Participants] — Participants were assessed for their PD-L1 tumor expression status by immunohistochemistry assay using archival tumor tissue or tumor tissue from a newly obtained biopsy. The PD-L1 tumor expression status of participants is presented. Population: All enrolled participants
  Participants
    Positive for PD-L1 | 53
    Negative for PD-L1 | 45
    Unknown PD-L1 Status | 5
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Count of Participants; unit: Participants] — Participants were assessed for ECOG PS: Grade 0: Fully active, able to carry on all pre-disease performance without restriction; Grade 1: Restricted in physically strenuous activity but ambulatory & able to carry out work of a light or sedentary nature; Grade 2: Ambulatory & capable of all selfcare but unable to carry out any work activities, up & about more than 50% of waking hours; Grade 3: Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; Grade 4: Completely disabled, cannot carry on any selfcare, totally confined to bed or chair or Grade 5: Dead. Population: All enrolled participants
  Participants
    ECOG PS=0 | 45
    ECOG PS=1 | 58
BRAF Mutation Expression Status [Count of Participants; unit: Participants] — BRAF mutation status was required from all participants. For participants that did not have a prior documented BRAF mutation status, BRAF V600 mutation analysis was performed by polymerase chain reaction (PCR) on tumor tissue. The BRAF mutation status of participants is presented. Population: All enrolled participants
  Participants
    Wild Type | 82
    Mutant | 20
    Unknown | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced At Least One Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a study treatment and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the study treatment or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that is temporally associated with the use of study treatment, is also an AE. The number of all participants who experienced at least one AE is presented.
Time Frame: Up to approximately 17 months (Through data cutoff date of 27-December-2017)
Population: The safety population consisted of all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Pembrolizumab: Participants received pembrolizumab 2 mg/kg IV on Day 1 of each 21-day cycle.
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 103
Participants | 101

2. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: The number of all participants who discontinued study treatment due to an AE is presented.
Time Frame: Up to approximately 17 months (through data cutoff date of 27-December-2017)
Population: The safety population consisted of all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 103
Participants | 4

3. Primary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: ORR was defined as the percentage of the participants in the analysis population who had a Complete Response (CR: disappearance of all target lesions) or a Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 assessed by blinded independent central review (BICR). The ORR per RECIST 1.1 for participants is presented. Participants without response data were treated as non-responders. ORR was analyzed using an exact method based on binomial distribution (Clopper-Pearson method) and is reported as percentage of participants.
Time Frame: Up to approximately 17 months (through data cutoff date of 27-December-2017)
Population: The analysis population consisted of all participants who received at least one dose of study treatment and had measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 102
Percentage of Participants | 16.7 [10.0 to 25.3]

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from first day of study treatment to death due to any cause. OS was analyzed using the Kaplan-Meier method and is reported in months.
Time Frame: Up to approximately 76 months
Population: The analysis population consisted of all participants who received at least one dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 103
Months | 13.2 [10.4 to 16.5]

5. Secondary Outcome: Progression-free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: PFS was defined as the time from the first day of study treatment to the first documented disease progression per RECIST 1.1 based on blinded independent central review (BICR) or death due to any cause, whichever occurred first. Using RECIST 1.1, progressive disease was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must have demonstrated an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered progression. PFS was analyzed using the Kaplan-Meier method and is reported in months. The PFS per RECIST 1.1 for participants is presented.
Time Frame: Up to approximately 76 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 102
Months | 2.8 [2.7 to 3.5]

6. Secondary Outcome: Duration of Response (DOR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: DOR was defined as the time from first documented evidence of Complete Response (CR: disappearance of all target lesions) or a Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 until disease progression or death due to any cause, whichever occurred first. Using RECIST 1.1, progressive disease was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must have demonstrated an absolute increase of at least 5 mm. DOR assessments were based on blinded independent central review (BICR). DOR was analyzed using the Kaplan-Meier method and is reported in months.
Time Frame: Up to approximately 76 months
Population: The analysis population consisted of all participants who received at least one dose of study treatment, had measurable disease at baseline, and had confirmed CR or PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 18
Months | 13.8 [5.5 to NA] — NA indicates upper limit of 95% CI for DOR cannot be calculated at the time of last disease assessment due to insufficient number of participants with response

7. Secondary Outcome: Objective Response Rate (ORR) Per Immune-related Response Evaluation Criteria in Solid Tumors (irRECIST)
Description: ORR was defined as the percentage of the participants in the analysis population who had a Complete Response (CR: disappearance of all lesions and no new lesions confirmed by a consecutive assessment at least 4 weeks after first documentation) or a Partial Response (PR: at least a 50% decrease in tumor burden relative to baseline confirmed by a consecutive assessment at least 4 weeks after first documentation) per irRECIST assessed by blinded independent central review (BICR). The ORR per irRECIST for participants is presented. Participants without response data were treated as non-responders. ORR was analyzed using an exact method based on binomial distribution (Clopper-Pearson method) and is reported as percentage of participants.
Time Frame: Up to approximately 76 months
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 102
Percentage of Participants | 18.6 [11.6 to 27.6]

8. Secondary Outcome: Progression-free Survival (PFS) Per Immune-related Response Evaluation Criteria in Solid Tumors (irRECIST)
Description: PFS was defined as the time from the first day of study treatment to the first documented disease progression per irRECIST based on blinded independent central review (BICR) or death due to any cause, whichever occurred first. Using irRECIST, progressive disease was defined as at least a 25% increase in tumor burden relative the minimum recorded tumor burden confirmed by a consecutive assessment at least 4 weeks after first documentation. PFS was analyzed using the Kaplan-Meier method and is reported in months. The PFS per irRECIST for participants is presented.
Time Frame: Up to approximately 76 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 102
Months | 2.8 [2.7 to 4.0]

9. Secondary Outcome: Duration of Response (DOR) by Immune-related Response Evaluation Criteria in Solid Tumors Version (irRECIST)
Description: DOR was defined as the time from first documented evidence of Complete Response (CR: disappearance of all lesions and no new lesions confirmed by a consecutive assessment at least 4 weeks after first documentation) or Partial Response (PR: at least a 50% decrease in tumor burden relative to baseline confirmed by a consecutive assessment at least 4 weeks after first documentation) per irRECIST until disease progression or death due to any cause, whichever occurred first. Using irRECIST, progressive disease was defined as at least a 25% increase in tumor burden relative the minimum recorded tumor burden confirmed by a consecutive assessment at least 4 weeks after first documentation. DOR assessments were based on blinded independent central review (BICR). DOR was analyzed using the Kaplan-Meier method and is reported in months.
Time Frame: Up to approximately 76 months
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 19
Months | 13.8 [5.4 to NA] — NA indicates upper limit of 95% CI for DOR cannot be calculated at the time of last disease assessment due to insufficient number of participants with response.

10. Secondary Outcome: Trough Serum Concentration (Ctrough) of Pembrolizumab Prior to Cycle 2 (21-day Cycle)
Description: Blood samples were obtained for PK analysis of the lowest (trough) concentration of pembrolizumab prior to the next dose of pembrolizumab administered during Cycle 2 (21-day cycle). The mean Ctrough of pembrolizumab prior to Cycle 2 is presented.
Time Frame: Day 21: Prior to the Cycle 2 (21-day cycle) Dose
Population: The analysis population consisted of participants who received 1 dose of study treatment, completed Cycle 1 (21-day cycle), and had blood samples drawn for Ctrough analysis.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 30
μg/mL | 8.70 (2.4)

11. Secondary Outcome: Trough Serum Concentration (Ctrough) of Pembrolizumab Prior to Cycle 4 (21-day Cycle)
Description: Blood samples were obtained for PK analysis of the lowest (trough) concentration of pembrolizumab prior to the next dose of pembrolizumab administered during Cycle 4 (21-day cycle). The mean Ctrough of pembrolizumab prior to Cycle 4 is presented.
Time Frame: Day 63: Prior to the Cycle 4 (21-day cycle) Dose
Population: The analysis population consisted of participants who received 3 doses of study treatment, completed Cycle 3 (21-day cycle), and had blood samples drawn for Ctrough analysis.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 26
μg/mL | 16.2 (6.7)

12. Secondary Outcome: Trough Serum Concentration (Ctrough) of Pembrolizumab Prior to Cycle 6 (21-day Cycle)
Description: Blood samples were obtained for PK analysis of the lowest (trough) concentration of pembrolizumab prior to the next dose of pembrolizumab administered during Cycle 6 (21-day cycle). The mean Ctrough of pembrolizumab prior to Cycle 6 is presented.
Time Frame: Day 105: Prior to the Cycle 6 (21-day cycle) Dose
Population: The analysis population consisted of participants who received 5 doses of study treatment, completed Cycle 5 (21-day cycle), and had blood samples drawn for Ctrough analysis.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 17
μg/mL | 22.9 (6.4)

13. Secondary Outcome: Trough Serum Concentration (Ctrough) of Pembrolizumab Prior to Cycle 8 (21-day Cycle)
Description: Blood samples were obtained for PK analysis of the lowest (trough) concentration of pembrolizumab prior to the next dose of pembrolizumab administered during Cycle 8 (21-day cycle). The mean Ctrough of pembrolizumab prior to Cycle 8 is presented.
Time Frame: Day 147: Prior to the Cycle 8 (21-day cycle) Dose
Population: The analysis population consisted of participants who received 7 doses of study treatment, completed Cycle 7 (21-day cycle), and had blood samples drawn for Ctrough analysis.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 13
μg/mL | 26.9 (6.5)

14. Secondary Outcome: Trough Serum Concentration (Ctrough) of Pembrolizumab Prior to Cycle 12 (21-day Cycle)
Description: Blood samples were obtained for PK analysis of the lowest (trough) concentration of pembrolizumab prior to the next dose of pembrolizumab administered during Cycle 12 (21-day cycle). The mean Ctrough of pembrolizumab prior to Cycle 12 is presented.
Time Frame: Day 231: Prior to the Cycle 12 (21-day cycle) Dose
Population: The analysis population consisted of participants who received 11 doses of study treatment, completed Cycle 11 (21-day cycle), and had blood samples drawn for Ctrough analysis.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 8
μg/mL | 33.8 (4.5)

15. Secondary Outcome: Trough Serum Concentration (Ctrough) of Pembrolizumab Prior to Cycle 16 (21-day Cycle)
Description: Blood samples were obtained for PK analysis of the lowest (trough) concentration of pembrolizumab prior to the next dose of pembrolizumab administered during Cycle 16 (21-day cycle). The mean Ctrough of pembrolizumab prior to Cycle 16 is presented.
Time Frame: Day 315: Prior to the Cycle 16 (21-day cycle) Dose
Population: The analysis population consisted of participants who received 15 doses of study treatment, completed Cycle 15 (21-day cycle), and had blood samples drawn for Ctrough analysis.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 4
μg/mL | 34.6 (5.0)

16. Secondary Outcome: Observed Maximum Serum Concentration (Cmax) of Pembrolizumab 30 Minutes After The End of Infusion During Cycle 1 (21-day Cycle)
Description: Blood samples were obtained for PK analysis of the Cmax of pembrolizumab 30 minutes after the end of infusion during Cycle 1 (21-day cycle). The Cmax of pembrolizumab is presented.
Time Frame: Day 0: 30 minutes after the end of infusion during Cycle 1 (21-day cycle)
Population: The analysis population consisted of participants who received 1 dose of study treatment in Cycle 1 (21-day cycle) and had blood samples drawn for Cmax analysis.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 28
μg/mL | 45.9 (10.9)

17. Secondary Outcome: Observed Maximum Serum Concentration (Cmax) of Pembrolizumab 30 Minutes After The End of Infusion During Cycle 8 (21-day Cycle)
Description: Blood samples were obtained for PK analysis of the Cmax of pembrolizumab 30 minutes after the end of infusion during Cycle 8 (21-day cycle). The Cmax of pembrolizumab is presented.
Time Frame: Day 147: 30 minutes after the end of infusion during Cycle 8 (21-day cycle)
Population: The analysis population consisted of participants who received 8 doses of study treatment and had blood samples drawn for Cmax analysis.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 12
μg/mL | 68.7 (12.5)

18. Secondary Outcome: Observed Serum Concentration of Pembrolizumab 1 Day After The End of Infusion During Cycle 1 (21-day Cycle)
Description: Blood samples were obtained for PK analysis of the serum concentration of pembrolizumab 1 day after the end of infusion during Cycle 1 (21-day cycle). The serum concentration of pembrolizumab is presented.
Time Frame: Day 2: 1 day after the end of infusion during Cycle 1 (21-day cycle)
Population: The analysis population consisted of participants who received 1 dose of study treatment in Cycle 1 (21-day cycle) and had blood samples drawn for serum concentration of pembrolizumab.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 30
μg/mL | 34.0 (4.6)

19. Secondary Outcome: Observed Serum Concentration of Pembrolizumab 5 Days After The End of Infusion During Cycle 1 (21-day Cycle)
Description: Blood samples were obtained for PK analysis of the serum concentration of pembrolizumab 5 days after the end of infusion during Cycle 1 (21-day cycle). The serum concentration of pembrolizumab is presented.
Time Frame: Day 6: 5 days after the end of infusion during Cycle 1 (21-day cycle)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 30
μg/mL | 18.4 (4.6)

20. Secondary Outcome: Observed Serum Concentration of Pembrolizumab 14 Days After The End of Infusion During Cycle 1 (21-day Cycle)
Description: Blood samples were obtained for PK analysis of the serum concentration of pembrolizumab 14 days after the end of infusion during Cycle 1 (21-day cycle). The serum concentration of pembrolizumab is presented.
Time Frame: Day 15: 14 days after the end of infusion during Cycle 1 (21-day cycle)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 30
μg/mL | 11.9 (2.5)

ADVERSE EVENTS:
Time Frame: Up to approximately 76 months.
Description: The safety population consisted of all participants who received at least one dose of study treatment. Per protocol, disease progression of cancer under study was not considered a serious AE (SAE) unless considered related to study treatment. Therefore, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study treatment are excluded as SAEs. One person who withdrew from the study (see participant flow) subsequently died.
Groups:
- Pembrolizumab Second Course: Eligible participants received up to 17 additional administrations (up to approximately 1 year) of pembrolizumab 2 mg/kg on day 1 of each 21-day cycle.
Arm/Group | Pembrolizumab | Pembrolizumab Second Course
All-Cause Mortality (participants affected / at risk) | 90/103 | 0/1
Serious Adverse Events (participants affected / at risk) | 13/103 | 0/1
Other Adverse Events (participants affected / at risk) | 98/103 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=103) | Pembrolizumab Second Course (N=1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Tumour rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=103) | Pembrolizumab Second Course (N=1)
Anaemia (Blood and lymphatic system disorders) | 27 (32) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 6 (6) | 0 (0)
Hypothyroidism (Endocrine disorders) | 27 (40) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 7 (7) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 7 (7) | 0 (0)
Constipation (Gastrointestinal disorders) | 8 (9) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 10 (12) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (8) | 1 (1)
Toothache (Gastrointestinal disorders) | 5 (5) | 1 (1)
Vomiting (Gastrointestinal disorders) | 11 (11) | 0 (0)
Asthenia (General disorders) | 8 (11) | 0 (0)
Fatigue (General disorders) | 16 (18) | 0 (0)
Pain (General disorders) | 7 (8) | 1 (1)
Pyrexia (General disorders) | 11 (14) | 0 (0)
Nasopharyngitis (Infections and infestations) | 6 (9) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 20 (25) | 0 (0)
Alanine aminotransferase increased (Investigations) | 28 (41) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 19 (29) | 0 (0)
Bilirubin conjugated increased (Investigations) | 11 (26) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 9 (10) | 0 (0)
Blood bilirubin increased (Investigations) | 19 (36) | 0 (0)
Blood bilirubin unconjugated increased (Investigations) | 7 (11) | 0 (0)
Blood cholesterol increased (Investigations) | 8 (16) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 12 (22) | 0 (0)
Blood glucose increased (Investigations) | 7 (9) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 17 (29) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (3)
Blood urea increased (Investigations) | 7 (11) | 0 (0)
Blood uric acid increased (Investigations) | 5 (14) | 1 (2)
Gamma-glutamyltransferase increased (Investigations) | 14 (17) | 0 (0)
Neutrophil count decreased (Investigations) | 11 (24) | 0 (0)
Platelet count increased (Investigations) | 6 (6) | 0 (0)
Total bile acids increased (Investigations) | 6 (13) | 0 (0)
Weight decreased (Investigations) | 14 (14) | 0 (0)
White blood cell count decreased (Investigations) | 13 (24) | 0 (0)
White blood cell count increased (Investigations) | 10 (13) | 0 (0)
White blood cells urine positive (Investigations) | 7 (8) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 19 (21) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 7 (14) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 12 (31) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 30 (67) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 14 (23) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 9 (11) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 9 (11) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (13) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (10) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 19 (25) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 1 (1)
Insomnia (Psychiatric disorders) | 9 (9) | 0 (0)
Proteinuria (Renal and urinary disorders) | 6 (6) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 16 (24) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 19 (20) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 15 (15) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-18): https://cdn.clinicaltrials.gov/large-docs/00/NCT02821000/Prot_SAP_001.pdf